CLINICAL TRIAL: NCT07149350
Title: Food Access, Value, and Optimization of Resources
Acronym: FAVORes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Allison Wu, Assistant Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00051793
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Food Insecurity; Health Behavior; Nutrition; Social Determinants of Health
Keywords: Nutrition Security; Food Insecurity; Group Coaching; Caregivers; Nutrition Education; Behavioral Intervention; Community-centered; Primary Care; Health-Related Social Needs; Food Access
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAVORes Workshop (Experimental): Participants will attend the FAVORes workshop, consisting of four weekly in-person group coaching sessions (1.5 hours each). Workshops are held at MEHC, led by a patient navigator, and are offered in English or in Spanish.
  Interventions: Behavioral: FAVORes Workshop

INTERVENTIONS:
Behavioral: FAVORes Workshop — The FAVORes (Food Access, Value, and Optimization of Resources) Workshop is a 4-week, in-person group coaching program for caregivers of children in food-insecure households. The intervention focuses on financial and nutrition literacy, community resource navigation, healthy eating habits, and setting family goals.

SUMMARY:
The main goal of the study is to examine the potential benefits of an educational workshop designed to help and support caregivers of children in families that struggle to get enough healthy food. The main questions are:

* Does the FAVORes workshop impact household food and nutrition security?
* Does the workshop change caregivers' knowledge, beliefs, and skills related to healthy food access?

Participants will:

* Attend four weekly in-person sessions (in English or Spanish)
* Complete short surveys
* Be interviewed after the workshop is completed (optional)

DETAILED DESCRIPTION:
The FAVORes (Food Access, Value, and Optimization of Resources) study at Boston Children's Martha Eliot Health Center (MEHC) aims to help families struggling with healthy food access. Over one in three families with children in Massachusetts face food insecurity. Further, they lack consistent access to nutritious food. Families face challenges such as insufficient knowledge of available resources, financial constraints, time scarcity, and/or language barriers. Social determinants such as food insecurity have adverse consequences on child health outcomes.

The FAVORes workshop is an in-person educational program for caregivers of children at MEHC. It is a 4-session, group coaching workshop led by a Senior Patient Navigator who shares her own experiences with food insecurity and as a health coach. The workshop runs over 4 weeks, 1.5 hours each session, is taught in small groups, and is available in both English and Spanish.

This workshop is designed to empower caregivers of children. It shares simple tips and steps to help with meal planning, having family meals, and eating healthier. The workshop also encourages caregivers to learn from each other in a group setting. Specific topics covered include setting "S.M.A.R.T. goals" (Specific, Measurable, Achievable, Relevant, Time-bound), understanding community food resources, managing time for healthy eating, and connecting food to overall health and mental well-being. The overall hypothesis for the FAVORes study is that the workshop will lead to meaningful and positive changes for families struggling with food insecurity.

Study Aims:

1. To examine the impact of the workshop on household food and nutrition security.
2. To explore changes in caregivers' knowledge, beliefs, and skills related to healthy food access.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Proficient in English or Spanish
* Attendance at the 1-hour "Towards Food Equity" Zoom session led by MEHC Social Work

Exclusion Criteria:

- Inability or anticipated inability to attend scheduled in-person workshop sessions for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-07 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Household Food Security Status at Baseline | At baseline (week 1)
  Mean score and proportion of participants classified by food security status based on the USDA Household Food Security Survey Module, 18-item version. Categorized by the raw score (0-18) into:
  Zero: High food security 1-2: Marginal food security 3-7: Low food security 8-18: Very low food security
Household Food Security Status at Week 4 | Week 4
  Mean score and proportion of participants classified by food security status based on the USDA Household Food Security Survey Module, 18-item version. Categorized by the raw score (0-18) into:
  Zero: High food security 1-2: Marginal food security 3-7: Low food security 8-18: Very low food security
Nutrition Security Status at Baseline | At baseline (week 1)
  Mean score and proportion of participants classified as nutrition secure/insecure using the 4-item nutrition security screener developed by the Center for Nutrition and Health Impact. Categorized by the raw score (0-4) into:
  0-2: Low nutrition security 3-4: High nutrition security
Nutrition Security Status at Week 4 | Week 4
  Mean score and proportion of participants classified as nutrition secure/insecure using the 4-item nutrition security screener developed by the Center for Nutrition and Health Impact. Categorized by the raw score (0-4) into:
  0-2: Low nutrition security 3-4: High nutrition security

SECONDARY OUTCOMES:
Participant reported confidence in setting S.M.A.R.T. goals at Week 4 | Week 4
  Proportion of participants responding "Agree" or "Strongly Agree" to the statement about increased confidence after the workshop, measured using a 5-point Likert scale: "After this workshop, I feel more confident in setting S.M.A.R.T. goals for my family."
Participant reported learning about new ways to make healthier food choices at Week 4 | Week 4
  Proportion of participants responding "Agree" or "Strongly Agree" to the statement about learning healthier food choices for their family, measured on a 5-point Likert scale: "I learned new ways to make healthier food choices for my family."
Participant reported knowledge about saving money on groceries in Week 4 | Week 4
  Proportion of participants reporting "Agree" or "Strongly Agree" to the ability to save money/use food budget better following the intervention, by Likert scale: "This workshop taught me how to save money on groceries and use my food budget better."
Participant reported knowledge of support programs/agencies in Week 4 | Week 4
  Proportion of participants reporting "Agree" or "Strongly Agree" to the statement about increased knowledge about agencies and programs available, by Likert scale: "I know more about programs and agencies that can help my family with food and other needs."
Participant reported improvement in family well-being in Week 4 | Week 4
  Proportion of participants reporting "Agree" or "Strongly Agree" to the statement: "Overall, this workshop has given me tools and knowledge to improve my family's well-being."
Participant reported workshop satisfaction in Week 4 | Week 4
  Proportion of participants reporting "Satisfied" or "Very Satisfied" with the workshop; measured via a 5-point satisfaction scale: "Overall, I am satisfied with my participation in the FAVORes workshop."
Participant reported likelihood of recommending workshop in Week 4 | Week 4
  Mean numeric score (0-10) for likelihood to recommend the workshop, using the Net Promoter Score question: "How likely are you to recommend this workshop to a friend or family member?" 0 = very unlikely, 5 = neutral, and 10 = extremely likely.

CONTACTS AND LOCATIONS:
Overall Officials: Allison J Wu, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Martha Eliot Health Center, Jamaica Plain, Massachusetts, United States